CLINICAL TRIAL: NCT03561259
Title: A Phase II, Open Label, Two-Arm Study of Therapeutic Iobenguane (131I) as Single Agent or in Combination With Vorinostat for Recurrent or Progressive High- Risk Neuroblastoma Subjects (OPTIMUM TRIAL)
Brief Title: A Study of Therapeutic Iobenguane (131-I) and Vorinostat for Recurrent or Progressive High-Risk Neuroblastoma Subjects
Acronym: OPTIMUM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jubilant DraxImage Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIBG 2014-01
Expanded Access: NCT01590680 (Available)
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Neuroblastoma; Neuroectodermal Tumors; Neoplasms
Keywords: Iobenguane Avid High-risk Neuroblastoma; 3-Iodobenzylguanidine; Radiopharmaceutical
MeSH Terms: conditions — Neuroblastoma; Neuroectodermal Tumors; Neoplasms | interventions — 3-Iodobenzylguanidine; Vorinostat

STUDY DESIGN:
Intervention Model Description: Two-arm, non-randomized, open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 131I-MIBG (Experimental): 131I-MIBG
  Interventions: Drug: 131I-MIBG
- 131I-MIBG + Vorinostat (Experimental): 131I-MIBG + Vorinostat
  Interventions: Drug: 131-MIBG + Vorinostat

INTERVENTIONS:
Drug: 131I-MIBG — Subjects will receive 18 mCi/kg of 131I-MIBG administered over 1.5 to 2 hours on Day 1 either a central line or a peripheral intravenous catheter. The maximum absolute dose of 131I-MIBG is determined by institution therapeutic limits and will not exceed 1,000 mCi. Subjects with an overall response of stable disease or better as assessed by the Investigator, and who meet certain protocol predefined criteria, may receive a second 18 mCi/kg 131I-MIBG treatment no sooner than 6 weeks following the first treatment.
  Other Names: I-131 meta-iodobenzylguanidine; Iobenguane I-131 MIBG Injection
  Arms: 131I-MIBG
Drug: 131-MIBG + Vorinostat — Subjects will receive vorinostat 180 mg/m2/dose (maximum dose 400 mg) once daily by mouth, NG, or G-tube on days -1 to +12 (14 total doses) for 14 days continuously. The 131I-MIBG treatment will be administered on day 1 via either a central line or a peripheral intravenous catheter over 1.5 to 2 hours. On day 1 of therapy, vorinostat should be taken 1 hour prior to the start of the 131I-MIBG infusion. Subjects with an overall response of stable disease or better, as assessed by the Investigator and who meet certain predefined criteria, may receive a second course of 18 mCi/kg 131I-MIBG combined with vorinostat (180 mg/m2) no sooner than 6 weeks following the first therapeutic 131I-MIBG treatment.
  Arms: 131I-MIBG + Vorinostat

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 131I-MIBG in combination with Vorinostat in patients with Recurrent or Progressive neuroblastoma

DETAILED DESCRIPTION:
OPTIMUM (MIBG 2014-01) is a Phase II, Two arm, non-randomized, open-label study of therapeutic 131I-iobenguane (131I-MIBG) as single agent or in combination with Vorinostat for the treatment of neuroblastoma. The study will be conducted in male and female subjects, greater than 1 year of age, with iobenguane avid, who have recurrent or progressive disease, regardless of overall response to frontline therapy, where frontline therapy includes a minimum of 4 cycles of induction therapy at any time prior to enrollment, high-risk neuroblastoma.

Subjects who are eligible for combination treatment will receive vorinostat 180 mg/m2/dose (maximum dose 400 mg) once daily for 14 days (Day -1 to Day 12) continuously.

Subjects will receive 18 mCi/kg of 131I-MIBG intravenously on Day 1.

If the subject qualifies, the subject will receive the second treatment course of 131I-MIBG in combination with vorinostat or 131I-MIBG alone (no sooner than 6 weeks following first treatment course). Subject must have an overall response of stable disease or better, as assessed by the Investigator, and meet certain predefined criteria to receive the second course of treatment.

Following a screening period of up to 4 weeks, the duration in the study treatment phase for an individual subject, who receives two treatments, is up to 26 weeks. For an individual subject, who receives one treatment only, the duration of the treatment phase is 16 weeks. In addition, there is a 2-year follow-up after the treatment phase, during which assessments will be performed to assess disease progression, as well as record adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a diagnosis of iobenguane avid, high-risk neuroblastoma based on Revised INRC criteria at the time of study enrollment with recurrent or progressive disease at any time prior to enrollment, regardless of overall response to frontline therapy, where frontline therapy includes a minimum of 4 cycles of induction therapy at any time prior to enrollment.
2. May have had prior 131I-MIBG therapy, provided:

   1. It has been at least 6 months from the date of last 131I-MIBG ;
   2. Response was other than progressive disease on first restaging after 131I-MIBG ;
   3. Prior 131I-MIBG was given as monotherapy and not in combination with systemic anticancer agents;
   4. Cumulative lifetime dose of 131I-MIBG at enrollment does not exceed 18 mCi/kg.
3. All soft tissue lesions identified on CT/MRI scans must be iobenguane avid lesions on an (123I)-iobenguane scan, or

   1. any progressive non-iobenguane avid lesion is proven by biopsy to be a non-neuroblastoma lesion.
   2. any other non-avid lesion is comprised of a fibrotic or scarred mass as shown by routine imaging and confirmed by the investigator.
4. Adequate cryopreserved autologous peripheral blood stem cells or bone marrow (at least 2 aliquots of 2.0 × 10exp6 CD34/kg at the time of study enrollment).
5. If a male, must agree to use an adequate contraception method as deemed appropriate by the Investigator (e.g., vasectomy, condoms) or partner using effective contraception and to not donate sperm during the study and for 90 days after receiving the last dose of study drug.
6. If a female of childbearing potential, have a negative serum pregnancy test result prior to each dosing and, if sexually active, be practicing an effective method of birth control [e.g., intrauterine device, double-barrier method (i.e., diaphragm, or a cervical cap) with intravaginal spermicidal foam, cream or gel], or male partner sterilization throughout the study.
7. Age at study entry ≥1 year.
8. Previous platelet transfusions are permitted, as long as the subject has a platelet count ≥50,000/μL without transfusion support for at least 1 week.
9. Subjects must have a minimum pulse oximetry measurement of at least 94% at baseline.
10. An absolute neutrophil count ≥750/μL without growth factor for 5 days.
11. Liver function parameter results: total bilirubin ≤2 × upper limit of normal for age, and Serum alanine aminotransferase (glutamic-pyruvic transaminase) and serum aspartate aminotransferase (glutamic-oxaloacetic transaminase) ≤ 10 times the upper limit of normal (for all sites, the upper limit of normal for alanine aminotransferase is defined as 45 U/L).
12. Normal thyroid function as measured by T4 or TSH or have abnormal results that are not considered clinically important by the Investigator or may be receiving levothyroxine.
13. Cardiac Function: shortening fraction of ≥ 27% by echocardiogram or ejection fraction ≥ 50% documented by echocardiogram or radionuclide angiogram within 1 month prior to Visit 1 (Baseline).
14. Karnofsky Performance Status (for subjects >16 years of age) or the Lansky Performance Status Performance Status (for subjects 1 to 16 years of age) ≥50%.
15. Full recovery from the toxic effects of any prior therapy.
16. Coagulation Function:

    1. International Normalized Ratio (INR) < 1.5
    2. Partial thromboplastin time (PTT) < 1.5 times upper limit of normal.

Exclusion Criteria:

1. Subjects within 5 half-lives after any antibody-based immunotherapy, or have not recovered from effects of any biologic therapy.
2. Subjects <12 weeks after myeloablative therapy with autologous stem cell transplant.
3. Subjects who have had an allogeneic stem cell treatment less than 4 months from Visit 1 are excluded. Those who have received allogeneic stem cell treatment more than 4 months from Visit 1 must have recovered and have no active graft versus host disease (GVHD) to be eligible.
4. Subjects must not have received radiation for a minimum of 2 weeks prior to study enrollment. Subjects whose only site(s) of disease have been radiated are eligible as long as the subject has MIBG avidity 2 weeks after completion of radiation. A minimum of 12 weeks prior to study enrollment is required following prior large field radiation therapy (ie, craniospinal, whole abdominal, total lung, > 50% marrow space)
5. History of total body irradiation.
6. Subjects do not have adequate renal function defined as GFR ≥ 70 mL/min/1.73 m2 either by creatinine clearance or radioisotope direct measurement or by calculation with the Schwartz formula
7. Subjects who are on hemodialysis.
8. Pregnancy or breastfeeding.
9. Significant active infections including active hepatitis B, or hepatitis C infection, or known infection with human immunodeficiency virus (HIV) (testing for HIV is not required prior to study entry).
10. Clinically important cardiac, pulmonary, and hepatic impairment.
11. Vorinostat treatment exclusion criteria (subjects, who meet any one of these criteria and otherwise meet eligibility criteria, are still eligible for 131I-MIBG monotherapy)

    1. Since valproic acid has HDAC inhibitory activity, patients must not have received valproic acid within 30 days of study entry.
    2. Since vorinostat may prolong the QT interval, patients must not be receiving other medications known to prolong the QT interval at the time of study entry . Pentamidine must not have been received within 1 week of study enrollment.
    3. Patients with a history of deep venous thrombosis that was not associated with the presence of a central venous catheter.
    4. Patients who are receiving Coumadin.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Overall Response | 6 weeks after the last 131I-MIBG treatment which will either be the first or the second treatment course (131I-MIBG + vorinostat) and a confirmatory assessment at least 6 weeks thereafter (at least 12 weeks from the end of treatment)
  Overall response (Yes/No) is based on the International Neuroblastoma Response Criteria (INRC, published 2017). The INRC will be calculated based on 123I-iobenguane scans, CT/MRI, and bone marrow biopsies and aspirates. A "Yes" is defined as complete response, partial response or minor response. A "No" response is defined as stable disease or progressive disease.

SECONDARY OUTCOMES:
Overall Response at 6 weeks after 131I-MIBG treatment | 6 weeks after the last 131I-MIBG treatment (first or second treatment of 131I-MIBG + vorinostat).
  The Revised INRC overall response (yes/no) defined as complete response, partial response, or minor response 6 weeks after the last131I-MIBG treatment which will either be the first treatment or the second treatment.
Durability of Effect of Overall Response (Yes/No) | For all tumour assessment data collected throughout the study (up to the end of the 2-year follow-up)(131I-MIBG + vorinostat).
  Durability of effect with the INRC will be assessed as INRC for all tumor assessment data available including any data collected beyond 12 weeks after the last 131I-MIBG treatment which will either be the first treatment or the second treatment.
Relative Curie Extension Score | 6 weeks after the last 131I-MIBG treatment which will either be the first or the second treatment course (131I-MIBG + vorinostat)
  Relative Curie Extension Score 6 weeks after the last MIBG 131I treatment, which will either be the first treatment or the second treatment.
Durability of Effect of Relative Curie Extension Score | For all tumour assessment data collected throughout the study for both arms (up to the end of the 2-year follow-up).
  Durability of effect with the Relative Curie Extension Score will be assessed as the score for all tumor assessment data available including any data collected beyond 12 weeks after the last MIBG 131I treatment, which will either be the first treatment or the second treatment. The Relative Curie Extension Score will be calculated using the Baseline (Visit 2) Absolute Curie Extension Score. The Curie Extension Scores will be calculated from the results of the (123I) iobenguane scans.

OTHER OUTCOMES:
Incidence of Adverse Events (CTCAE Version 5.0) | Up to 22 weeks
  Adverse events as graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Incidence of Serious Adverse Events | Through study completion, up to 2.5 years.
  Percentage of subjects with hematological and nonhematological toxicities. Any relationship between the whole body radiation absorbed dose and nonhematological SAEs will also be assessed;
Whole Body Radiation Dose | After each 131I-MIBG treatment for up to 120 hours.
  To assess radiation safety in terms of any potential relationship between the whole body radiation absorbed dose and nonhematological serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Melda Dolan, Study Director — Jubilant DraxImage Inc., dba Jubilant Radiopharma
Locations (21):
- United States (21):
  - Stanford University, Palo Alto, California
  - UCSF Pediatric Hematology/Oncology, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University Medical Center in St. Louis, St Louis, Missouri
  - Northwell Health /Cohen Children's Medical Center, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Children's Hospital (Atrium Health), Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Children's Health, Dallas, Texas
  - Cook Children's Hematology/Oncology Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin, American Family Children's Hospital and Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No